CLINICAL TRIAL: NCT01011348
Title: Q10 for Gulf War Veterans
Acronym: GULF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: W81WH-07-1-0667
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Gulf War Illness
Keywords: Gulf War Illness; Coenzyme Q10; Quality of Life; Fatigue; oxidative stress
MeSH Terms: conditions — Fatigue | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo vs Q10 100mg vs Q10 300mg (Other)
  Interventions: Dietary Supplement: Coenzyme Q10; Dietary Supplement: Placebo
- Q10 100mg vs Placebo vs Q10 300mg (Other)
  Interventions: Dietary Supplement: Coenzyme Q10; Dietary Supplement: Placebo
- Placebo vs. Q10 300mg vs. Q10 100mg (Other)
  Interventions: Dietary Supplement: Coenzyme Q10; Dietary Supplement: Placebo
- Q10 300mg vs. Placebo vs. Q10 100mg (Other)
  Interventions: Dietary Supplement: Coenzyme Q10; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — 100mg/day for three months
  Other Names: PharmaNord Myoquinione softgel caplets
Dietary Supplement: Coenzyme Q10 — 300mg/day for three months
  Other Names: PharmaNord Myoquinione softgel caplets
Dietary Supplement: Placebo — Three month period
  Other Names: PharmaNord matched identical softgel placebo

SUMMARY:
Goal: The investigators propose to test whether giving the supplement coenzyme Q10 (Q10) improves symptoms and subjective health in Gulf War veterans (GWV) with chronic, multi-symptom health problems.

Rationale: Direct empirical evidence, in groups that are not GWV, has supported benefit of Q10 to many of the symptoms that GWV are at heightened risk of experiencing - such as fatigue, muscle pain, and cognition, which are syndrome-defining conditions. In addition, Q10 has also been reported to benefit other symptoms arising at increased rates in GWV, including headaches, sleep disturbances, and breathing problems. This provides a strong rationale for testing whether Q10 will have similar benefit to these symptoms in GWV.

Method: 46 GWV with chronic health problems will participate.The design is a randomized, double-blind, placebo-controlled crossover study. Each subject will be "crossed over" between Q10 and an identical placebo, receiving each agent twice, for 3.5 month periods. In one of the Q10 phases, a lower dose of Q10 will be used - 100mg three times a day; while in one a higher dose will be used - 300mg three times a day. Neither subjects nor investigators will know which substance each subject is receiving in which phase. Subjects will be randomly assigned to one of four crossover orders.

Assessments: Assessments will include subjective quality of life; symptoms that are "syndrome defining" for Gulf War illness (like fatigue and muscle problems); and other symptoms and conditions reported to occur more commonly in GWV (like sleep problems). Analyses will show whether Q10 led to improvements when compared to placebo; whether higher Q10 doses improved outcomes more than lower doses; and whether people with certain symptoms or characteristics get more benefit than people with other symptoms or characteristics.

DETAILED DESCRIPTION:
Goal: To determine, via a double-blind placebo-controlled crossover study, whether coenzyme Q10 (Q10) administration reduces symptoms and improve subjective health in Gulf War veterans (GWV).

Rationale: In a number of settings, studies have reported benefits of Q10 to fatigue, muscle pain and cognition, "syndrome" defining symptoms in GWV. It has also been reported to improve a range of other symptoms and conditions that arise at increased rates in GWV. Additionally Q10 defends against mechanisms that may play a role in health problems in GWV. For these reasons, a study evaluating benefits by Q10 to symptoms and quality of life in symptomatic GWV is merited.

Subjects: 46 GWV meeting Center for Disease Control (CDC) and Kansas criteria for "Gulf War illness." Design: Randomized, placebo-controlled, double-blind crossover study. Intervention: Coenzyme Q10 at 100mg three times a day (tid) or 300mg tid or matching placebo for 3.5 ± 0.5 month periods.

Primary Outcome: Subjective health; syndrome defining symptoms (fatigue, muscle pain, muscle strength; and cognition).

Secondary Outcomes: A variety of secondary outcomes will be assessed including other symptoms reported to be elevated in GWV; markers of oxidative stress; and dose-response.

Analyses: Nonparametric and secondarily parametric analyses will compare effects of Q10 vs placebo; and of higher dose vs lower dose Q10 on primary and secondary endpoints. Possible effect modification (differential benefit) based on factors such as oxidative state and Q10 serum concentration will be explored through regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Deployed to the Middle East for any period between August 1990 and July 1991.
* Adherence to CDC criteria for Gulf War illness: Chronic symptoms, for at least six months, first arising after Gulf deployment, in at least two of the three areas of fatigue, musculoskeletal, and mood/cognition.
* Adherence to Kansas criteria for Gulf War illness. To aid specificity, these criteria are more involved than CDC criteria Veterans are asked about symptoms in several general categories (e.g., respiratory, gastrointestinal, neuropsychological, sleep disturbances, pain), as well as symptoms (e.g., fatigue, headache) for which no single category is apparent. Gulf War illness criteria symptoms must have persisted or recurred in the year prior to interview and first have been a problem for respondents in 1990 or later. Full criteria are as delineated in Steele 2000.
* Willing to agree to defer initiating other over the counter medications till after completion of study participation.
* Willing to defer participation in other clinical trials till after completion of study participation.
* If female of childbearing potential, willing to be on two forms of birth control during study participation.

Exclusion Criteria:

* Any factor that might compromise participation for the full duration of the study.
* Known active cancer (except nonmelanoma skin cancer), neurodegenerative disease, or HIV.
* Active medical problems distinct from Gulf War symptomatology that confer a significant probability of hospitalization, medication change, or change in clinical state during the course of participation.
* Use of coumadin.
* Use of Q10-containing products, including lotions, toothpastes, or supplements in the prior two months.
* Current use of drugs known to be mitochondrial toxins: amiodarone, protease inhibitors, fluoroquinoline ("floxin") antibiotics.
* Nursing or pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Coenzyme Q10 will improve overall subjective quality of life in ill Gulf War Veterans, using a single item General Self-Rated Health measure. | Assessed every three months for one year

SECONDARY OUTCOMES:
Coenzyme Q10 will improve specific symptoms that dominate definitions of illness in GWV including fatigue, pain, and muscle strength. | Assessed every three months over one year
Coenzyme Q10 will subjectively improve other symptoms reported to arise at elevated rates in GWV defined by responses on a symptom survey (e.g. headache, shortness of breath, sleep problems, gastrointestinal problems). | Assessed every three months over one year
Effect modification: The magnitude of Coenzyme Q10 (Q10) benefit may be influenced by baseline oxidative state, change in oxidation with Q10, and serum Q10 level; or by which symptoms a veteran has. | Assessed every three months over one year
Assess whether higher dose Q10 provides greater benefit; or does so selectively in individuals with more unfavorable baseline oxidation state; or individuals who require a higher dose to achieve the same change in Q10, e.g. due to impaired assimilation. | Assessed every three months over one year

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice A Golomb, M.D., Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Erickson LC, Ritchie JB, Javors JM, Golomb BA. Recruiting a special sample with sparse resources: lessons from a study of Gulf War veterans. Clin Trials. 2013;10(3):473-82. doi: 10.1177/1740774512470040. Epub 2013 Jan 16. PMID 23325028